CLINICAL TRIAL: NCT00722371
Title: A Multicenter, Randomized, Double-Blind Study of the Co-Administration of Sitagliptin and Pioglitazone in Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control
Brief Title: MK0431 and Pioglitazone Co-Administration Factorial Study in Patients With Type 2 Diabetes Mellitus (0431-102 AM2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-102; 2008_522 (Other: Merck Study Number)
Record Dates: First submitted 2008-07-22; First posted 2008-07-25 (Estimated); Results first posted 2011-10-17 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Pioglitazone; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- Sitagliptin 100 mg (Experimental)
  Interventions: Drug: Sitagliptin phosphate; Drug: Matching placebo to pioglitazone; Drug: Metformin
- Pioglitazone 15 mg (Experimental)
  Interventions: Drug: Pioglitazone hydrochloride; Drug: Matching placebo to sitagliptin; Drug: Metformin
- Pioglitazone 30 mg (Experimental)
  Interventions: Drug: Pioglitazone hydrochloride; Drug: Matching placebo to sitagliptin; Drug: Metformin
- Pioglitazone 45 mg (Experimental)
  Interventions: Drug: Pioglitazone hydrochloride; Drug: Matching placebo to sitagliptin; Drug: Metformin
- Sitagliptin 100 mg/ Pioglitazone 15 mg (Experimental)
  Interventions: Drug: Sitagliptin phosphate; Drug: Pioglitazone hydrochloride; Drug: Metformin
- Sitagliptin 100 mg/ Pioglitazone 30 mg (Experimental)
  Interventions: Drug: Sitagliptin phosphate; Drug: Pioglitazone hydrochloride; Drug: Metformin
- Sitagliptin 100 mg/ Pioglitazone 45 mg (Experimental)
  Interventions: Drug: Sitagliptin phosphate; Drug: Pioglitazone hydrochloride; Drug: Metformin

INTERVENTIONS:
Drug: Sitagliptin phosphate — Sitagliptin 100 mg tablet (blinded) orally once daily for 54 weeks.
  Other Names: Januvia; Tesavel; Xelevia; Ristaben
  Arms: Sitagliptin 100 mg; Sitagliptin 100 mg/ Pioglitazone 15 mg; Sitagliptin 100 mg/ Pioglitazone 30 mg; Sitagliptin 100 mg/ Pioglitazone 45 mg
Drug: Pioglitazone hydrochloride — Pioglitazone 15 mg, 30 mg, or 45 mg tablets or capsules (blinded) orally once daily for 54 weeks. Participants randomized to receive pioglitazone 45 mg as monotherapy or in combination with sitagliptin were to start on pioglitazone 30 mg at Week 1 and undergo uptitration to pioglitazone 45 mg at Week 4.
  Other Names: Actos
  Arms: Pioglitazone 15 mg; Pioglitazone 30 mg; Pioglitazone 45 mg; Sitagliptin 100 mg/ Pioglitazone 15 mg; Sitagliptin 100 mg/ Pioglitazone 30 mg; Sitagliptin 100 mg/ Pioglitazone 45 mg
Drug: Matching placebo to sitagliptin — Matching placebo to sitagliptin orally once daily for 54 weeks.
  Arms: Pioglitazone 15 mg; Pioglitazone 30 mg; Pioglitazone 45 mg
Drug: Matching placebo to pioglitazone — Matching placebo to pioglitazone tablets or capsules orally once daily for 54 weeks.
  Arms: Sitagliptin 100 mg
Drug: Metformin — Metformin 500 mg (open-label) was to be initiated as rescue therapy to participants not meeting specific glycemic goals. The dose of metformin may have been uptitrated and adjusted, at the discretion of the investigator, up to the maximum approved dose in the country of origin.

SUMMARY:
A study to evaluate the efficacy and safety of sitagliptin and pioglitazone co-administration in comparison with sitagliptin and pioglitazone monotherapy in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Patient is highly unlikely to conceive
* Patient meets one of the 3 categories is naïve to all antihyperglycemic agent (AHA) therapies, or is non-naïve based upon the patient's current diet, medical regimen and screening A1c patient is currently not on AHA with a screening A1c >=7.5 % and =<11.0 % patient is currently on either metformin pr sulfonylurea monotherapy with a screening A1c >=7.0 % and =<9.0 %

Exclusion Criteria

* Patient has a history of type 1 diabetes mellitus or history of ketoacidosis or has C=peptide value of =<0.8 ng/mL
* Patient has previously been treated with insulin, thiazolidinedione (TZD) (rosiglitazone or pioglitazone), any Dipeptidyl peptidase-4 (DPP-4) inhibitor (sitagliptin, vildagliptin, or alogliptin), exenatide or has previously been in a clinical study with any DPP-4 inhibitor or incretin mimetic
* Patient is on a weight loss program and is not in the maintenance phase or has started a weight loss medication (e.g. orlistat or sibutramine) within the prior 8 weeks
* Patient has undergone surgery within the prior 30 days or has major surgery planned during the study
* Patient has a medical history of active liver disease including chronic active hepatitis B or C or symptomatic gallbladder disease including primary biliary cirrhosis
* Patient has received treatment with an investigational product within 12 weeks prior to Visit 1

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1615 (Actual)
Dates: Start 2008-09-05 (Actual); Primary Completion 2010-10-26 (Actual); Study Completion 2011-03-25 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Henry RR, Staels B, Fonseca VA, Chou MZ, Teng R, Golm GT, Langdon RB, Kaufman KD, Steinberg H, Goldstein BJ. Efficacy and safety of initial combination treatment with sitagliptin and pioglitazone--a factorial study. Diabetes Obes Metab. 2014 Mar;16(3):223-30. doi: 10.1111/dom.12194. Epub 2013 Aug 29. PMID 23909985

RESULTS

PARTICIPANT FLOW:
Groups:
- Sitagliptin 100 mg: Sitagliptin 100 mg and matching placebo to pioglitazone once daily for 54 weeks.
- Pioglitazone 15 mg: Pioglitazone 15 mg and matching placebo to sitagliptin once daily for 54 weeks.
- Pioglitazone 30 mg: Pioglitazone 30 mg and matching placebo to sitagliptin once daily for 54 weeks.
- Pioglitazone 45 mg: Pioglitazone 45 mg and matching placebo to sitagliptin once daily for 54 weeks.
- Sitagliptin 100 mg/ Pioglitazone 15 mg: Sitagliptin 100 mg and pioglitazone 15 mg once daily for 54 weeks.
- Sitagliptin 100 mg/ Pioglitazone 30 mg: Sitagliptin 100 mg and pioglitazone 30 mg once daily for 54 weeks.
- Sitagliptin 100 mg/ Pioglitazone 45 mg: Sitagliptin 100 mg and pioglitazone 45 mg once daily for 54 weeks.
Period: Overall Study
Arm/Group | Sitagliptin 100 mg | Pioglitazone 15 mg | Pioglitazone 30 mg | Pioglitazone 45 mg | Sitagliptin 100 mg/ Pioglitazone 15 mg | Sitagliptin 100 mg/ Pioglitazone 30 mg | Sitagliptin 100 mg/ Pioglitazone 45 mg
Started | 231 | 230 | 233 | 230 | 230 | 231 | 230
Completed | 175 | 158 | 168 | 167 | 182 | 178 | 179
Not Completed | 56 | 72 | 65 | 63 | 48 | 53 | 51
Not completed — Adverse Event | 6 | 13 | 9 | 10 | 6 | 8 | 4
Not completed — Contraindication | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Creatinine / Creatinine clearance | 2 | 1 | 2 | 3 | 2 | 1 | 1
Not completed — Excluded medication | 0 | 1 | 1 | 0 | 0 | 0 | 1
Not completed — Hyperglycemia | 2 | 6 | 4 | 2 | 5 | 1 | 1
Not completed — Hypoglycemia | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 4 | 6 | 6 | 6 | 2 | 3 | 0
Not completed — Lost to Follow-up | 11 | 14 | 21 | 13 | 8 | 16 | 13
Not completed — Physician Decision | 5 | 2 | 2 | 5 | 2 | 3 | 4
Not completed — Pregnancy | 1 | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 6 | 1 | 0 | 1 | 4 | 2 | 1
Not completed — Withdrawal by Subject | 18 | 27 | 19 | 23 | 19 | 18 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin 100 mg | Pioglitazone 15 mg | Pioglitazone 30 mg | Pioglitazone 45 mg | Sitagliptin 100 mg/ Pioglitazone 15 mg | Sitagliptin 100 mg/ Pioglitazone 30 mg | Sitagliptin 100 mg/ Pioglitazone 45 mg | Total
Number analyzed (Participants) | 231 | 230 | 233 | 230 | 230 | 231 | 230 | 1615
Age, Customized [Number; unit: Participants]
  <=20 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  21 to 30 years | 5 | 6 | 2 | 5 | 5 | 8 | 4 | 35
  31 to 40 years | 37 | 39 | 33 | 20 | 17 | 34 | 15 | 195
  41 to 50 years | 64 | 73 | 60 | 70 | 73 | 60 | 68 | 468
  51 to 60 years | 83 | 67 | 88 | 76 | 80 | 75 | 87 | 556
  61 to 70 years | 31 | 34 | 45 | 53 | 44 | 49 | 51 | 307
  >70 years | 11 | 11 | 5 | 6 | 11 | 5 | 5 | 54
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 82 | 106 | 117 | 112 | 96 | 95 | 703
  Male | 136 | 148 | 127 | 113 | 118 | 135 | 135 | 912

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1C (A1C) at Week 24
Description: A1C represents the percentage of glycosylated hemoglobin.
Time Frame: Baseline and Week 24
Population: Full Analysis Set with last observation carried forward (LOCF). Reasons for exclusion included no baseline data and/or no post-baseline data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of glycosylated hemoglobin
Arm/Group | Sitagliptin 100 mg | Pioglitazone 15 mg | Pioglitazone 30 mg | Pioglitazone 45 mg | Sitagliptin 100 mg/ Pioglitazone 15 mg | Sitagliptin 100 mg/ Pioglitazone 30 mg | Sitagliptin 100 mg/ Pioglitazone 45 mg
Number analyzed (Participants) | 172 | 163 | 181 | 171 | 179 | 173 | 188
Percentage of glycosylated hemoglobin | -1.09 [-1.29 to -0.89] | -0.88 [-1.09 to -0.68] | -1.21 [-1.41 to -1.02] | -1.20 [-1.40 to -1.00] | -1.53 [-1.73 to -1.34] | -1.63 [-1.82 to -1.43] | -1.81 [-2.00 to -1.62]

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24
Time Frame: Baseline and Week 24
Population: Full Analysis Set with LOCF. Reasons for exclusion included no baseline data and/or no post-baseline data.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin 100 mg | Pioglitazone 15 mg | Pioglitazone 30 mg | Pioglitazone 45 mg | Sitagliptin 100 mg/ Pioglitazone 15 mg | Sitagliptin 100 mg/ Pioglitazone 30 mg | Sitagliptin 100 mg/ Pioglitazone 45 mg
Number analyzed (Participants) | 179 | 176 | 185 | 181 | 189 | 181 | 193
mg/dL | -24.3 [-32.0 to -16.5] | -19.5 [-27.2 to -11.7] | -29.9 [-37.6 to -22.3] | -37.4 [-45.1 to -29.7] | -41.0 [-48.5 to -33.5] | -46.9 [-54.6 to -39.3] | -52.0 [-59.6 to -44.5]

3. Secondary Outcome: Change From Baseline in 2-Hour Post-meal Glucose (PMG) at Week 24
Description: PMG was measured using the Meal Tolerance Test (MTT).
Time Frame: Baseline and Week 24
Population: Full Analysis Set with LOCF. Reasons for exclusion included no baseline data and/or no post-baseline data.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin 100 mg | Pioglitazone 15 mg | Pioglitazone 30 mg | Pioglitazone 45 mg | Sitagliptin 100 mg/ Pioglitazone 15 mg | Sitagliptin 100 mg/ Pioglitazone 30 mg | Sitagliptin 100 mg/ Pioglitazone 45 mg
Number analyzed (Participants) | 141 | 128 | 158 | 136 | 149 | 143 | 154
mg/dL | -51.1 [-64.0 to -38.2] | -30.6 [-44.0 to -17.3] | -52.5 [-64.9 to -40.2] | -66.6 [-79.8 to -53.5] | -69.2 [-81.7 to -56.7] | -85.5 [-98.4 to -72.6] | -93.8 [-106.4 to -81.2]

4. Primary Outcome: Change From Baseline in A1C at Week 54
Description: A1C represents the percentage of glycosylated hemoglobin.
Time Frame: Baseline and Week 54
Population: Full Analysis Set with LOCF. Reasons for exclusion included no baseline data and/or no post-baseline data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent of glycosylated hemoglobin
Arm/Group | Sitagliptin 100 mg | Pioglitazone 15 mg | Pioglitazone 30 mg | Pioglitazone 45 mg | Sitagliptin 100 mg/ Pioglitazone 15 mg | Sitagliptin 100 mg/ Pioglitazone 30 mg | Sitagliptin 100 mg/ Pioglitazone 45 mg
Number analyzed (Participants) | 172 | 163 | 181 | 171 | 179 | 173 | 188
Percent of glycosylated hemoglobin | -0.93 [-1.15 to -0.72] | -0.74 [-0.96 to -0.53] | -1.16 [-1.37 to -0.95] | -1.23 [-1.45 to -1.02] | -1.45 [-1.65 to -1.24] | -1.49 [-1.71 to -1.28] | -1.78 [-1.99 to -1.58]

5. Secondary Outcome: Change From Baseline in FPG at Week 54
Time Frame: Baseline and Week 54
Population: Full Analysis Set with LOCF. Reasons for exclusion included no baseline data and/or no post-baseline data.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin 100 mg | Pioglitazone 15 mg | Pioglitazone 30 mg | Pioglitazone 45 mg | Sitagliptin 100 mg/ Pioglitazone 15 mg | Sitagliptin 100 mg/ Pioglitazone 30 mg | Sitagliptin 100 mg/ Pioglitazone 45 mg
Number analyzed (Participants) | 179 | 176 | 185 | 181 | 189 | 181 | 193
mg/dL | -13.1 [-21.6 to -4.5] | -10.5 [-19.0 to -2.0] | -24.0 [-32.4 to -15.5] | -33.3 [-41.8 to -24.8] | -33.9 [-42.2 to -25.7] | -37.1 [-45.5 to -28.6] | -47.8 [-56.1 to -39.5]

6. Secondary Outcome: Change From Baseline in 2-Hour PMG at Week 54
Description: PMG was measured using the Meal Tolerance Test (MTT).
Time Frame: Baseline and Week 54
Population: Full Analysis Set with LOCF. Reasons for exclusion included no baseline data and/or no post-baseline data.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin 100 mg | Pioglitazone 15 mg | Pioglitazone 30 mg | Pioglitazone 45 mg | Sitagliptin 100 mg/ Pioglitazone 15 mg | Sitagliptin 100 mg/ Pioglitazone 30 mg | Sitagliptin 100 mg/ Pioglitazone 45 mg
Number analyzed (Participants) | 145 | 131 | 158 | 141 | 150 | 143 | 157
mg/dL | -37.0 [-50.2 to -23.7] | -26.7 [-40.5 to -13.0] | -46.8 [-59.6 to -34.1] | -58.2 [-71.6 to -44.7] | -64.7 [-77.6 to -51.8] | -69.7 [-83.1 to -56.4] | -88.2 [-101.2 to -75.3]

ADVERSE EVENTS:
Arm/Group | Sitagliptin 100 mg | Pioglitazone 15 mg | Pioglitazone 30 mg | Pioglitazone 45 mg | Sitagliptin 100 mg/ Pioglitazone 15 mg | Sitagliptin 100 mg/ Pioglitazone 30 mg | Sitagliptin 100 mg/ Pioglitazone 45 mg
Serious Adverse Events (participants affected / at risk) | 14/231 | 10/230 | 5/233 | 11/230 | 12/230 | 15/231 | 7/230
Other Adverse Events (participants affected / at risk) | 60/231 | 41/230 | 45/233 | 55/230 | 48/230 | 56/231 | 46/230
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin 100 mg (N=231) | Pioglitazone 15 mg (N=230) | Pioglitazone 30 mg (N=233) | Pioglitazone 45 mg (N=230) | Sitagliptin 100 mg/ Pioglitazone 15 mg (N=230) | Sitagliptin 100 mg/ Pioglitazone 30 mg (N=231) | Sitagliptin 100 mg/ Pioglitazone 45 mg (N=230)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mitral valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Optic ischaemic neuropathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dengue fever (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Splenic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Prostate cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Complicated migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin 100 mg (N=231) | Pioglitazone 15 mg (N=230) | Pioglitazone 30 mg (N=233) | Pioglitazone 45 mg (N=230) | Sitagliptin 100 mg/ Pioglitazone 15 mg (N=230) | Sitagliptin 100 mg/ Pioglitazone 30 mg (N=231) | Sitagliptin 100 mg/ Pioglitazone 45 mg (N=230)
Nasopharyngitis (Infections and infestations) | 13 (13) | 10 (11) | 12 (16) | 9 (10) | 12 (15) | 15 (19) | 8 (10)
Upper respiratory tract infection (Infections and infestations) | 10 (13) | 6 (6) | 8 (9) | 12 (12) | 11 (13) | 9 (11) | 11 (13)
Hypoglycaemia (Metabolism and nutrition disorders) | 25 (57) | 20 (30) | 22 (78) | 20 (81) | 20 (45) | 26 (100) | 24 (93)
Headache (Nervous system disorders) | 17 (18) | 6 (8) | 9 (9) | 11 (12) | 8 (8) | 14 (18) | 5 (5)
Hypertension (Vascular disorders) | 7 (8) | 5 (5) | 4 (4) | 10 (11) | 13 (13) | 6 (9) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation.